CLINICAL TRIAL: NCT03543631
Title: Survey on Precision Medicine and Digital Health
Acronym: precisionmed
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Shelly Meese, Admin, Project Manager (not PI), Scripps Health
Other Study IDs: precision_medicine
Record Dates: First submitted 2018-05-03; First posted 2018-06-01 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Health Behavior; Health Knowledge, Attitudes, Practice; Health Attitude
MeSH Terms: conditions — Health Behavior; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Online survey

SUMMARY:
The investigators have created an anonymous online survey that queries current topics in precision medicine.

DETAILED DESCRIPTION:
The investigators have created an anonymous online survey to assess the educational requirements and current gaps in knowledge related to advances in precision medicine. These include questions that focus on digital health, wearable technologies, genetic sequencing, and CRISPR to assess survey participants' interest and knowledge level.

ELIGIBILITY:
Inclusion Criteria:

* Students and physicians at all levels of training.

Exclusion Criteria:

* None.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone who access and is interested in participating in the online survey.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Precision medicine | August 2018 - November 2018
  To assess survey participants' knowledge of precision medicine using multiple choice methodologies.

SECONDARY OUTCOMES:
Digital health | August 2018 - November 2018
  To determine whether participants use a health monitoring device from multiple choice methodologies.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Bi, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No